CLINICAL TRIAL: NCT05162053
Title: A Phase 1, Open-label, Randomized, Multiple-dose, Crossover Pharmacokinetic/Pharmacodynamic Study of Vicagrel and Clopidogrel in Healthy Subjects With Different CYP2C19 Phenotypes
Brief Title: PK/PD Study of Vicagrel and Clopidogrel in Healthy Subjects With Different CYP2C19 Metabolizers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VCP1-Ⅰ-06
Record Dates: First submitted 2021-12-14; First posted 2021-12-17 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — methyl 2-(2-acetoxy-6,7-dihydrothieno(3,2-c)pyridin-5(4H)-yl)-2-(2-chlorophenyl)acetate; Clopidogrel

STUDY DESIGN:
Intervention Model Description: Multiple-center, open-label, randomized, multiple-dose, crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ultra-rapid metabolizers group (Experimental): A 7-day cross-dosing of vicagrel and clopidogrel between two cycles
  Interventions: Drug: vicagrel Capsules; Drug: Clopidogrel Tablets
- Rapid metabolizers group (Experimental): A 7-day cross-dosing of vicagrel and clopidogrel between two cycles
  Interventions: Drug: vicagrel Capsules; Drug: Clopidogrel Tablets
- Normal metabolizers group (Experimental): A 7-day cross-dosing of vicagrel and clopidogrel between two cycles
  Interventions: Drug: vicagrel Capsules; Drug: Clopidogrel Tablets
- Intermediate metabolizers group (Experimental): A 7-day cross-dosing of vicagrel and clopidogrel between two cycles
  Interventions: Drug: vicagrel Capsules; Drug: Clopidogrel Tablets
- Poor metabolizers group (Experimental): A 7-day cross-dosing of vicagrel and clopidogrel between two cycles
  Interventions: Drug: vicagrel Capsules; Drug: Clopidogrel Tablets

INTERVENTIONS:
Drug: vicagrel Capsules — Oral administration for 7 days under fasting
Drug: Clopidogrel Tablets — Oral administration for 7 days under fasting
  Other Names: PLAVIX

SUMMARY:
This clinical study will adopt an open-label, randomized, multiple-dose, two-crossover design to explore the pharmacokinetic and pharmacodynamic profiles of Vicagrel Capsules and Clopidogrel Tablets in Healthy Subjects with Different CYP2C19 Metabolizers

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent before study, and fully understand the study content, process and possible adverse reactions;
2. Able to complete the study in compliance with the protocol;
3. Subject (including partner) is willing to voluntarily take effective contraceptive measures from screening through 90 days after the last dose of study drug (see Appendix 5 for details);
4. Male and female subjects between the ages of 18 and 65 years, inclusive;
5. At least 50 kg for male subjects, 45 kg for female subjects, with a Body Mass Index (BMI= Weight/Height2) between 18-32 kg/m2, inclusive;
6. With normal or clinically insignificant abnormal results of physical examination and vital signs test;
7. Subjects will be assigned into the group according to the CYP2C19 genotype: the first group of ultra-rapid metabolizers (CYP2C19*17/*17); the second group of rapid metabolizers (CYP2C19*1/*17); the third group of normal metabolizers (CYP2C19*1/*1); the fourth group of intermediate metabolizers (CYP2C19*1/*2, *1/*3, *2/*17, *3/*17); and the fifth group of poor metabolizers (CYP2C19*2/*2, *2/*3, *3/*3).。

Exclusion Criteria:

1. More than 5 cigarettes per day on average within 3 months before the study;
2. History of sensitivity to drugs similar to the study drug or have high sensitivity to clopidogrel, allergic constitution (e.g. allergy to various drugs and foods);
3. History of drug abuse, drug use, alcohol abuse (14 units of alcohol per week: 1 units = 285 mL beer, 25 mL spirit or 100 mL wines);
4. Donation or loss of a significant volume of blood (> 450 mL) within 56 days prior to screening;
5. Intake of any prescription drugs, over-the-counter drugs, vitamin or herbal medicine within 14 days prior to receiving study drug;
6. Consumption of any special diet (such as grapefruit, pitaya, mango, pomelo, etc.) or subjects have engaged strenuous exercise or any other factors affecting drug absorption, distribution, metabolism and excretion within 14 days prior to receiving study drug;
7. Intake of any drug which Have taken strong inhibitors and/or inducers of liver metabolic enzymes (CYP1A2, 2A6, 2C8, 2C19, 3A4 and 3A5) within 28 days before the first medication, and strong inhibitors of liver metabolic enzymes such as: ciprofloxacin, clopidogrel, Itraconazole, ketoconazole, ritonavir, troleandomycin, etc., strong inducers of liver metabolism enzymes such as: rifampicin, carbamazepine, phenytoin sodium, St. John's wort, etc.(For details see Appendix 6);
8. Recent major changes in diet or exercise habits;
9. Use of an investigational drug or product, or participation in a drug research study within 30 days (or 5 half-lives) prior to receiving study drug;
10. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption;
11. Suffering from any diseases that may increase the risk of bleeding, such as hemorrhoids, acute gastritis, stomach and duodenal ulcers, Thrombocytopenic Purpura and hemophilia, etc;
12. Family history of coagulation or bleeding disorders (e.g., hemophilia)/symptoms (e.g., vomiting blood, black stools, severe or recurrent nosebleeds, coughing up blood, significant hematuria, or intracranial hemorrhage) or suspected vascular malformations, such as aneurysms or early onset strokes, in the individual or in their immediate family;
13. A clinically significant 12-lead ECG abnormality;
14. Positive test results of blood pregnancy or subject is lactating for female subjects;
15. Any clinically significant abnormalities/findings in laboratory tests, or any clinically significant disease including but not limited to gastrointestinal, renal, hepatic, neurological system, blood, endocrine, tumor, lung, immune, mental, or cardiovascular and cerebrovascular diseases;
16. Positive test results for viral hepatitis (including hepatitis B and C), HIV antibody or syphilis antibody;
17. Acute illness or concomitant medication from screening to the first dosing of study medication;
18. Consumption of chocolate or any food or beverages containing caffeine or (rich containing) xanthine within 48 h prior to receiving the first dosing of study medication;
19. Consumption of any product containing alcohol within 24 h prior to receiving the first dosing of study medication, or positive results from a screen for alcohol;
20. Positive results from a screen for urine drug test (Morphine, marijuana);
21. Subjects were vaccinated within 4 weeks prior to screening, or planned to be vaccinated during the trial;
22. Any condition which in the opinion of Investigator is not suitable for subjects to participate in the study (For ultra-rapid metabolizers and rapid metabolizers, investigators may consider at their discretion).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Inhibition of platelet aggregation [IPA] evaluated in healthy subjects to treatment with either vicagrel or clopidogrel | Day1-Day31
  To compare IPA following multiple doses of vicagrel and/or clopidogrel in healthy subjects with different CYP2C19 phenotypes.
Platelet reactivity index [PRI] evaluated in healthy subjects to treatment with either vicagrel or clopidogrel | Day1-Day31
  To compare PRI following multiple doses of vicagrel and/or clopidogrel in healthy subjects with different CYP2C19 phenotypes.
maximum plasma concentration (Cmax) | Day1-Day31
  To compare Cmax following multiple doses of vicagrel and/or clopidogrel in healthy subjects with different CYP2C19 phenotypes.
Area under the curve over a dosing interval(AUC0-tau) | Day1-Day31
  To compare AUC0-tau following multiple doses of vicagrel and/or clopidogrel in healthy subjects with different CYP2C19 phenotypes.

SECONDARY OUTCOMES:
Assess the safety and tolerability of multiple doses of both drugs in each CYP2C19 phenotype group. | Day1-Day31

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Principal Investigator — Phase I Clinical Research Center of The First Hospital of Jilin University; Youngjun David Kim, MD, Principal Investigator — Altasciences Clinical, Los Angeles; Martin Kankam, MD, Principal Investigator — Altasciences, Kansas City
Locations (3):
- United States (2):
  - Altasciences Clinical, Los Angeles, Los Angeles, California
  - Altasciences, Kansas City, Kansas City, Missouri
- Phase I Clinical Research Center of The First Hospital of Jilin University, Changchun, Jilin, China